CLINICAL TRIAL: NCT04257370
Title: An Open Label, Randomized Controlled Study to Compare Healing of Severe Diabetic Foot Ulcers and Forefoot Amputations in Diabetics With and Without Moderate Peripheral Arterial Disease Treated With Kerecis Omega3 Wound and SOC vs. SOC Alone
Brief Title: Kerecis Omega3 Wound Plus SOC vs. SOC Alone in Treating Severe Diabetic Foot Ulcers and Forefoot Amputations
Acronym: Odinn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Collaborators: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other); Allderma Pharmaceuticals (Unknown); Endospin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS-0370
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Foot Ulcer; Dehiscence of Amputation Stump; Amputation
Keywords: Diabetic foot ulcer; DFU; Dehisced amputation; Acute amputation; Fish skin; Kerecis
MeSH Terms: conditions — Diabetic Foot; Ichthyosis Vulgaris | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to receive either Kerecis™ Omega3 Wound plus standard of care, or standard or care alone.
Who Masked: Outcomes Assessor
Masking Description: Evaluation of wound closure at defined time points will be done by an assessor blinded to the treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kerecis™ Omega3 Wound (Experimental)
  Interventions: Device: Kerecis™ Omega3 Wound
- Standard of care (Active Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Kerecis™ Omega3 Wound — Kerecis™ Omega3 Wound is decellularised, intact fish skin from North Atlantic cod fish. Kerecis™ Omega3 Wound is FDA approved and EU cleared for the treatment of diabetic ulcers, chronic vascular ulcers, venous ulcers, trauma wounds (including abrasions, lacerations, and skin tears), acute surgical wounds (including debridement, amputation, and donor sites), surgical wounds (dehiscence or failed healing after surgery), imminent failure of STSG, and post-injection necrosis.
  Arms: Kerecis™ Omega3 Wound
Other: Standard of care — Standard of care wound treatment as defined by the local site, including debridement of the wound, standard wound dressing, and proper offloading of the wound site.
  Arms: Standard of care

SUMMARY:
This is a prospective, multi-national, multi-centre, randomized, non-blinded (photo evaluation is blinded), controlled clinical investigation in patients suffering from diabetic wounds reaching to tendon, bone, or joint. Patients will be randomised to received intact fish skin (Kerecis™ Omega3 Wound) plus standard of care or standard of care alone, and wound healing compared over 16 weeks.

DETAILED DESCRIPTION:
This study is a multi-center study in France, Germany, Italy, and Sweden on the healing effect of Kerecis™ Omega3 Wound in severe diabetic ulcers and open amputation wounds compared to standard of care treatment.

Cell and/or tissue based wound treatment products (CTPs) have been advancing in the treatment of non-healing ulcers in the last 20 years. In 2013, a new product was approved in Europe and by the FDA, intact fish skin, delivered as a sterilized, freeze-dried material, for the treatment of acute and chronic wounds. Fish skin has the benefit of not requiring treatment with antibiotics, or virus inactivating methods, thereby allowing the natural content of the skin to remain, and is a by-product of food industry. Therefore, the fish derived CTP is both ecologically sustainable as well as rich in naturally occurring soluble molecules and omega-3 fatty acids.

A study evaluating the prognosis of diabetic ulcers from large registry data found that the deeper, larger, and more long-standing ulcers would take longer to heal. If a wound was older than 2 months, larger than 2 cm2 and reached bone or tendon, the likelihood of healing in 20 weeks was 19%. The average cost to close a diabetic foot wound with advanced moist wound healing has been calculated at €2300 per cm2, so closing a 3 cm2 wound would cost €6900..

A wealth of clinical experience on diabetic wounds exists on the Kerecis fish skin material. This is, however, mainly in the form of case series and has been published through posters and case reports. The main indication for Kerecis is deep or non-healing diabetic ulcers, which are the biggest problem in diabetic wound care ultimately leading to amputation. Studies on CTPs have almost solely been done on shallow diabetic ulcers to get a homogeneous study population which then is randomized to treatment with the studied product or the control product. This means that in the case of a favourable outcome in the study, those products are not really tested on the ulcer for which they are ultimately intended, ulcers where the next step is amputation.

This randomized controlled study on deep diabetic wounds is designed to prove the efficacy of Kerecis™ Omega3 Wound for the indications it is intended for - severe diabetic foot ulcers - and to show the cost effectiveness of using Kerecis™ Omega3 Wound over standard of care. Wounds resulting from an amputation that are left open with an opening into bone, or from a dehisced amputation where the sutures have gone up, are included. Acute amputations where the metatarsal bones are exposed are included, provided that the patient has diabetes and the amputation is a result of an ulcer.

This study is probably the first study on severe diabetic ulcers where the CTP is used on the types of wounds that it is intended for, thereby giving a straight answer to the actual savings included in healing a serious diabetic wound earlier or changing the stage to a smaller shallower ulcer (changing grade of ulcer), thus, radically changing the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient with chronic lower extremity wounds: Grade 2 or 3 according to University of Texas score: Grade 2: "Wounds that penetrate to tendon or capsule". Grade 3: "wounds that penetrate to bone or into the joint". In this context, probing gently to bone means that the wound reaches bone.
* OR patients with diabetes that are recently amputated below the ankle, where the wound has not been closed or has dehisced and bones/tendons are exposed.
* Patients that have moderately decreased or normal arterial circulation. In this study the cutoff point is Ankle Brachial Index (ABP) below 0.6. (Toe pressure and TPCO2 values will be obtained if possible. Toe pressure of 50mmHg and a TCPO2 value of 40mm on the dorsum of the foot is often considered as indicative of adequate perfusion.)
* Patients who will tolerate aggressive debridement. Light bleeding of the wound surface should be seen after debridement.
* Patient has had his/her ulcer for one month.
* Participant is willing and able to give informed consent for participation in the clinical trial.
* Male or Female, over 18 years.
* Geographical distance compatible with taking part in the study. Observe though that the patient can be treated at a "home clinic" every other week as long as the end point is not imminent and photos and acetate tracers with cm markers are fed into the photo portal.
* Negative pregnancy test for a woman of childbearing age.
* Patient is able (in the investigator's opinion) and willing to comply with all the clinical trial requirements.

Exclusion Criteria:

* Patient whose wound surface is not measurable.
* Patients suffering from unmanaged osteomyelitis. With adequate treatment the patient can be re-screened for the study.
* Patient with severe ischemia (Ankle Brachial Index (ABI) <0.6).
* Patient with necrotic wound who will not tolerate aggressive debridement.
* Patient with immune deficiency or autoimmune disease.
* Patients having done arterial reconstruction within one month. These patients can be re-screened later.
* Patient on systemic corticosteroids or other treatments causing delayed wound healing.
* Female participants who are pregnant, breast feeding or planning pregnancy during the course of the clinical trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the clinical trial, or may influence the result of the clinical trial, or the participant's ability to participate in the clinical trial.
* Patient with known allergy to fish.
* Patient deprived of liberty by judicial or administrative decision, person subject to a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Wound healing at Week 16 | 16 weeks
  Percentage of patients with complete wound epithelialisation at 16 weeks as assessed from photographs by a blinded assessor

SECONDARY OUTCOMES:
Ulcer grade | 16 weeks
  Change in grade of ulcer according to the University of Texas diabetic wound classification at each weekly visit
Change in quality of life | 16 weeks
  Change in quality of life as assessed by a Wound Quality of Life questionnaire at each weekly visit. The questionnaire contains 17 questions about the patients' wounds and patients will be asked to rate between five values (e.g. Does your wound hurt? Available answers: "not at all", "a little", "moderately", "quite a lot", and "very much").
Change in pain | 16 weeks
  Pain will be assessed by a visual analogue scale (VAS) at each weekly visit. The VAS will range from 0-10, with 0 being no pain at all, and 10 being worst pain imaginable, and patients will be asked to self-evaluate the pain they experience.
Healing trajectory | 16 weeks
  Healing trajectories will be plotted via the change in wound surface area in cm2, vs original wound size, calculated at each weekly visit
Cost effectiveness | 16 weeks
  Better cost-effectiveness than standard of care as calculated by global cost of wound treatment of the two arms and projected costs for non-healed ulcers
Number of participants with fully healed ulcers at 20 weeks | 20 weeks
  The number of patients with wounds with complete epithelialisation at 20 weeks will be calculated for each arm (checkpoint only)
Number of participants with fully healed ulcers at 24 weeks | 24 weeks
  The number of patients with wounds with complete epithelialisation at 24 weeks will be calculated for each arm (checkpoint only)
Percentage of ulcers healed 50% or more at 12 weeks | 12 weeks
  The percentage of ulcers healed 50% or more at 12 weeks will be compared between groups. 50% healing indicates epithelialisation of 50% of the original wound area in cm2.

CONTACTS AND LOCATIONS:
Overall Officials: Dured Dardari, MD, PhD, Principal Investigator — CHSF
Locations (1):
- Centre Hospitalier Sud Francilien, Évry, Corbeil-Essonnes Cedex, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margolis DJ, Allen-Taylor L, Hoffstad O, Berlin JA. Diabetic neuropathic foot ulcers: predicting which ones will not heal. Am J Med. 2003 Dec 1;115(8):627-31. doi: 10.1016/j.amjmed.2003.06.006. PMID 14656615
- [Background] Barshes NR, Sigireddi M, Wrobel JS, Mahankali A, Robbins JM, Kougias P, Armstrong DG. The system of care for the diabetic foot: objectives, outcomes, and opportunities. Diabet Foot Ankle. 2013 Oct 10;4. doi: 10.3402/dfa.v4i0.21847. PMID 24130936
- [Derived] Dardari D, Piaggesi A, Potier L, Sultan A, Diener H, Francois M, Dorweiler B, Bouillet B, M'Bemba J, Chaillous L, Clerici G, Kessler L, Wetzel-Roth W, Storck M, Davidsson OB, Baldursson B, Kjartansson H, Lantis JC, Charpentier G. Intact Fish Skin Graft to Treat Deep Diabetic Foot Ulcers. NEJM Evid. 2024 Dec;3(12):EVIDoa2400171. doi: 10.1056/EVIDoa2400171. Epub 2024 Oct 4. PMID 39365895